CLINICAL TRIAL: NCT06265896
Title: Effect of Kinesiotaping on Activation of Abdominal Muscles in Female Patients With Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Nagy Mamdouh, Principal Investigator (M.Sc. student), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004948
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Kinesiotaping; Abdominal Muscles; Female Patients; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping +Pelvic floor exercise training (Experimental): They will be treated by Elastic Kinesio-tape of (K-Active) brand which will be applied over abdomen, which will be changed every 3 days and this will be maintained along four weeks, plus conventional pelvic floor exercises; 30 minutes, 3 times/week for 12 sessions.
  Interventions: Other: Kinesio taping; Other: Pelvic floor exercise training
- Pelvic floor exercise training (Active Comparator): They will be treated by conventional pelvic floor exercises; 30 minutes, 3 times/week for 12 sessions.
  Interventions: Other: Pelvic floor exercise training

INTERVENTIONS:
Other: Kinesio taping — Tape will be applied on rectus abdominis muscles using muscles facilitation technique from origin to insertion of muscle with a tension between 15-35%. Band will start on symphysis pubis with no tension and then women make stretch on the abdominal region by deep abdominal inspiration and will end at xiphoid process. Tape will be applied on the right and left external oblique muscles; the procedure will start without tension from bottom and of 6-12 ribs, then the hip will be placed in flexion and rotation to opposite direction and the tape will be attached to pubic bone with tension between 15-35%. Finally, the tape will be performed on the right and left internal oblique muscles; the procedure will start without tension from anterior superior iliac spine and then the hip will be placed in extension position and the tape will be attached to lower 4 ribs and linea alba with tension between 15-35%.
  Arms: Kinesio taping +Pelvic floor exercise training
Other: Pelvic floor exercise training — The intervention will be applied by a trained physical therapist. First of all, each participant will be instructed to relax thighs, bottom and abdomen musculature, then squeeze pelvic floor muscles 'focus on tightening without flexing abdomen, thighs or buttocks- avoid holding breath' 10 repetitions, 3 to 5 times a day (morning, afternoon, and night). Rest for 4 seconds and then repeat each contraction. Build up pelvic floor musculatures strength until each participant be able to do 10 slow contractions each time, holding them for 10 seconds each with rests of 4 seconds in between. Then do not hold your breath or tighten your stomach, bottom or thigh muscles at the same time. Will instruct participants to try holding each squeeze for a few seconds.

SUMMARY:
This study will be conducted to evaluate the effect of kinesiotaping on activation of abdominopelvic cavity for management of stress urinary incontinence females' patients.

DETAILED DESCRIPTION:
Stress urinary incontinence, the involuntary leakage of urine during exercise or certain movements, is a common pelvic floor disorder that can negatively impact quality of life. Urinary incontinence is associated with reduced physical, social, and mental well-being. While alternative exercise regimens have been proposed, It was concluded there is insufficient evidence they reduce leakage in women with stress urinary incontinence.

Kinesio taping is a rehabilitative technique that provides support and stability to muscles using elastic tape. Kinesio tape has no drugs/chemicals and allows normal skin function.

Limited studies have shown taping specific abdominal areas can stimulate skin-organ reflexes and improve pelvic organ function through interactions between the pelvis, pelvic floor muscles, and synergists. Therefore, could suggested that KT application on abdominopelvic cavity might be emerged as a conservative treatment option for urinary incontinence There were couple of previous research investigated the KT efficacy on treating bladder over activity with promising results of improvements. Till now, there is no previous study illustrating the effect of kinesio taping on abdominopelvic cavity in stress urinary incontinence females. So, this study will be the first one in this issue. Therefore, it will have valuable benefits in physical therapy field and scientific research.

ELIGIBILITY:
Inclusion Criteria:

1. Women suffering from mild to moderate stress urinary incontinence, clinically diagnosed by the gynecologist.
2. Their ages will be ranged from 30-50 years old.
3. Their body mass index (BMI) will be ranged from (20-25 kg/m2).
4. They shouldn't have any musculoskeletal or neurological disorders.

Exclusion Criteria:

1. Current pregnancy.
2. Malignant condition
3. History of acute infection
4. Neurological problem
5. Mental problem to prevent evaluation and cooperation
6. Having allergies to kinesiotaping
7. Having uncontrolled metabolic diseases like diabetes and thyroid disease.
8. Athletic females

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor impact questionnaire- short form 7 (PFIQ-7) | 4 weeks
  It will be used to evaluate the efficacy of a particular therapy, and to compare bladder, bowel or vaginal symptoms severity for all females in both groups (A&B) before and after treatment. All of the items use the following response scale: 0, Not at all; 1, somewhat; 2, moderately; 3, quite a bit PFIQ-7 Score, Obtain the mean value for all of the answered items within the corresponding scale (possible value 0- 3) and then multiply by (100/3) to obtain the scale score (range 0-100). The final score is the sum of the scores from the 3 scales together to obtain the summary score (range 0-300).
King's Health Questionnaire (KHQ) | 4 weeks
  The KHQ is a validated instrument for measuring the quality of life of women with urinary incontinence. This questionnaire consists of two parts and 32 items. The first part (21 items) contains two single-item questions that address General Health Perception and Incontinence Impact and the following seven multi-item domains: Role, Physical, and Social Limitations, Limitations in Personal Relationship, Emotional Problems, Sleep and Energy Disturbances associated with SUI, and Severity Measures for UI. The second part has an 11-item Symptom Severity Scale (SSS) that assesses the presence and severity of urinary symptoms. While the entire SSS is scored from 0 (best) to 30 (worst), the minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health) for all other KHQ domains.

SECONDARY OUTCOMES:
Assessment of pelvic floor muscle strength | 4 weeks
  The pelvic floor muscle strength will be assessed using a perineometer for all females in both groups (A&B) before and after treatment. Each participant will be positioned relaxed in supine with flexed, slightly abducted legs, where each participant will be asked to insert the probe that will be covered by condom and be lubricated with hypoallergic gel into her vaginal cavity, where 0.5-1 centimeter of the probe sustained visible outside of her introitus. Then each participant will be asked to squeeze by a maximum voluntary contraction in three repetitions, each will be last by 3 seconds, with 3 seconds rest in-between, Then, a 2-minutes rest break will be taken, followed by visible contraction of transversus abdominis muscle, as long without pelvic tilting. And will take the median of the three measures.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia M. Kamel, Prof., Study Chair — Department of Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Cairo University, Giza, Egypt